CLINICAL TRIAL: NCT02011737
Title: The Effectiveness and Safety of Naftopidil 75mg for Improving Clearance of Ureteral and Renal Stones After Shockwave Lithotripsy: Prospective Randomized Controlled Study
Brief Title: Naftopidil 75mg for Improving Clearance of Urinary Stones
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Principal Investigator, HAN, DEOK HYUN, Assistant Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMC2013-08-066
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Kidney Calculi; Ureter Calculi
Keywords: Medical Expulsive therapy
MeSH Terms: conditions — Kidney Calculi | interventions — naftopidil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naftopidil (Active Comparator): Naftopidil 75mg once daily
  Interventions: Drug: naftopidil 75mg
- Placebo (Placebo Comparator): Placebo once daily

INTERVENTIONS:
Drug: naftopidil 75mg
  Arms: Naftopidil

SUMMARY:
The purpose of this study is to evaluate Efficacy and Safety of oral intake of Naftopidil 75mg once daily for the improving clearance of ureteral or renal stones.

DETAILED DESCRIPTION:
Prospective, Single-center, Double blind, Randomized controlled trial

Treatment

- Oral Naftopidil 75 mg once daily are given to the patients who are scheduled for shockwave lithotripsy (ESWL) because of ureteral or renal stones.

Follow up Assessments including X-ray(KUB), visual analogue pain scale, are done 2, 4, and 6 weeks after the ESWL.

ELIGIBILITY:
Inclusion Criteria:

* Radio-opaque (identifiable in KUB) ureter or kidney calculi
* size criteria is from 5mm to 15mm

Exclusion Criteria:

* Symptomatic acute urinary tract infection during the run-in period
* severe hydronephrosis
* 2 or more urinary stones
* Radiolucent (non-visible in KUB) stone
* recent intervention for the urinary stone within 6 month
* Patients who have ureteral stent
* over 2.0 mg/dl of serum creatinine level
* severe hepatic dysfunction
* orthostatic hypotension
* current usage of alpha-adrenergic blocker or calcium channel blocker
* Pregnant or nursing women
* Age under 15 year
* severe or uncontrolled medical conditions

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Difference of the treatment success rate in two weeks after ESWL between treatment group and placebo group | 2 weeks after ESWL
  Treatment success is defined as no or less than 3 mm size remnant stone

SECONDARY OUTCOMES:
Difference of the treatment success rate after ESWL between treatment group and placebo group | 4, 6 weeks after ESWL
  Treatment success is defined as no or less than 3 mm size remnant stone
Adverse Event | 2,4,6weeks
  Rate of total Adverse Events and Adverse Events relevant to Investigational drug
pain scale | baseline, 2, 4, 6 weeks
  visual analogue pain scale due to urinary stone
rate of additional intervention | 6 week
  incidence of additional intervention for the urinary stone ex> ureteral stent insertion, percutaneous nephrostomy, ureteroscopic ureterolithotomy, percutaneous nephrolithotomy, laparoscopic stone removal and so on

OTHER OUTCOMES:
time to stone expulsion | 2,4,6week
  the time (days) elapsed from first ESWL to the expulsion of the stone
Number of ESWL | 6week
  The number of required ESWL for the stone expulsion

CONTACTS AND LOCATIONS:
Overall Officials: Deok Hyun Han, M.D., Principal Investigator — Department of Urology, Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Seoul, South Korea